CLINICAL TRIAL: NCT00759629
Title: An International, Multicenter, Randomized Trial Assessing the Value of Mechanical Reperfusion in Patients With Acute Myocardial Infarction Presenting > 12 Hours From Onset of Symptoms
Brief Title: Beyond 12 Hours Reperfusion AlternatiVe Evaluation Trial
Acronym: Brave-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. I00800
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Interventional treatment group - Patients assigned to PCI will receive the loading dose of clopidogrel, aspirin plus a bolus of heparin and be transferred immediately for interventional treatment. They will receive abciximab as a bolus followed by a continuous infusion of for 12 hours.
  Interventions: Other: Interventional treatment group
- B (Active Comparator): Conservative treatment group - Patients assigned to this group will receive the usual therapy in the intensive care unit of the admitting hospital according to local standards.
  Interventions: Other: Conservative treatment group

INTERVENTIONS:
Other: Interventional treatment group — Patients assigned to PCI will receive the loading dose of clopidogrel (300 mg), 500 mg aspirin plus a bolus of 70 U/kg heparin i.v. and be transferred immediately for interventional treatment. They will receive abciximab as a bolus of 0.25 mg/Kg of body weight followed by a continuous infusion of 0.125 µg/Kg/minute (up to a maximal dose of 10 µg/minute) for 12 hours. All patients will undergo coronary angiography and left ventriculography in the conventional way. During the procedure patients will receive the weight-adjusted heparin doses (70 U/ kg). Post-procedural antithrombotic therapy will consist of clopidogrel in a daily dose of 75 mg for at least 4 weeks (6 months recommended) and aspirin, 100 mg to 350 mg daily, indefinitely.
  Arms: A
Other: Conservative treatment group — Patients assigned to this group will receive the usual therapy in the intensive care unit of the admitting hospital according to local standards. Per protocol, all patients in this arm will receive a loading dose of clopidogrel (300 mg) followed by 75 mg/day for at least 4 weeks (6 months recommended) after randomization and aspirin, indefinitely. Recommended additional regimen will include heparin, ß-blockers, ACE inhibitors and statins
  Arms: B

SUMMARY:
The objective of this international, multicenter, randomized study is to assess whether coronary artery stenting is associated with a reduced infarct size in patients with AMI presenting between 12 and 48 hours after onset of symptoms compared to medical treatment alone

DETAILED DESCRIPTION:
Between 8.5% and 40% of patients with acute myocardial infarction present late after symptom onset, no longer being eligible for thrombolysis.Despite efforts to reduce time to presentation, recent studies have demonstrated that time-to-arrival has not changed.The lack of efficacy of thrombolysis in patients with acute MI presenting > 12 hours after symptom onset may be a reason why current guidelines oppose reperfusion therapy in this setting.Several findings suggest, however,that reperfusion therapy may be beneficial even among these patients. First, recent studies have shown that viable salvageable myocardium exists even after >12 hours of severe ischemia. Second, previous studies have not only demonstrated that PCI is better than thrombolysis in patients with acute MI,but also that the time window of efficacy for PCI may be wider than that for thrombolysis.Third, observational studies suggest that PCI is effective even when performed after 12 hours from symptom onset in patients with acute MI. The goal of our trial was to assess whether an invasive strategy based on PCI with stenting is associated with reduction of infarct size in patients with acute STEMI presenting > 12 hours after symptom onset compared with a conventional conservative treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilling the criteria of AMI and presenting at the hospital between 12 and 48 hours after onset of symptoms. The criteria of AMI are fulfilled when at least one episode of typical chest pain lasting ≥ 20 minutes is combined with either unequivocal ECG changes (≥ 0.1 mV of ST-segment elevation in ≥ 2 limb leads or ≥ 0.2 mV in ≥ 2 contiguous precordial leads or new pathological Q-waves) or CK plus concomitant CK-MB increase above twice the upper normal threshold. All patients have to be informed of the nature of the study and should give their informed consent for participation in the study.

Exclusion Criteria:

* Age <18 years and > 80 years
* Cardiogenic shock (systolic blood pressure < 80 mm Hg unresponsive to fluids or necessitating the infusion of catecholamines: GUSTO I criteria)
* Persistent severe chest pain
* Prior thrombolysis (for index AMI)
* Malignancies with life expectancy < 1year
* History of bleeding diathesis, coagulopathy
* Contraindications to the antithrombotic therapy used in conjunction with coronary stenting (clopidogrel and abciximab)
* Stroke within the past 3 months
* Major surgery within the past 30 days
* Platelets < 100000/mm3 or >700000/mm3, Hb < 10g/dl, white blood cell count <3000/mm3
* Percutaneous coronary intervention within the past 30 days
* Inability to cooperate with study procedures and/or follow-up
* Previous enrollment in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2001-05; Primary Completion 2005-01 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the infarct size calculated as the final perfusion defect (% of left ventricle) at the scintigraphic study | 5-10 days

SECONDARY OUTCOMES:
Secondary endpoint of the study is the composite of all-cause death, recurrent MI, or stroke within 30 days after randomization. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schoemig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (14):
- Landeskrankenhaus Feldkirch, Feldkirch, Austria
- Germany (11):
  - Staedtisches Krankenhaus Bad Reichenhall, Bad Reichenhall
  - Kreiskrankenhaus Erding/Dorfen, Erding
  - Kreiskrankenhaus Freilassing, Freilassing
  - Kreisklinik Fuerstenfeldbruck, Fürstenfeldbruck
  - Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - Deutsches Herzzentrum Muenchen, Munich
  - 1st Medizinische Klinik, Klinikum rechts der Isar, Munich
  - Krankenhaus Vinzentinum Ruhpolding, Ruhpolding
  - Krankenhaus Schongau, Schongau
  - Klinikum Traunstein, Traunstein
  - Kreisklinik Trostberg, Trostberg an der Alz
- Italy (2):
  - Azienda Ospedaliera Careggi, Florence
  - Ospedale, "Umberto I", Mestre

REFERENCES:
- [Result] Schomig A, Mehilli J, Antoniucci D, Ndrepepa G, Markwardt C, Di Pede F, Nekolla SG, Schlotterbeck K, Schuhlen H, Pache J, Seyfarth M, Martinoff S, Benzer W, Schmitt C, Dirschinger J, Schwaiger M, Kastrati A; Beyond 12 hours Reperfusion AlternatiVe Evaluation (BRAVE-2) Trial Investigators. Mechanical reperfusion in patients with acute myocardial infarction presenting more than 12 hours from symptom onset: a randomized controlled trial. JAMA. 2005 Jun 15;293(23):2865-72. doi: 10.1001/jama.293.23.2865. PMID 15956631